CLINICAL TRIAL: NCT02811315
Title: Flutiform Treatment in Patients With Asthma in Daily Clinical Practice; a Prospective Observational Non-interventional Study Assessing the Effect of Space Use and Adherence on Fluticasone/Formoterol FDC Efficacy Measured With the Asthma Control Questionnaire (ACQ-6).
Brief Title: Flutiform in Treatment of Patients With Asthma in Daily Clinical Practice.
Status: Withdrawn | Type: Observational
Why Stopped: Lack of interest
Sponsor: Mundipharma Pharmaceuticals B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: FLT9509
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational. Non interventional study — Observational. Non interventional study

SUMMARY:
The objective of the study is to evaluate the effect of frequency of use with a spacer on asthma control in Dutch patients with asthma during their daily clinical practice over 12 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to be prescribed fluticasone/formoterol fixed dose combination as follows:

Patients not adequately controlled in inhaled corticosteriods and "as required" inhaled short acting beta 2 agonist or patients already adequately controlled on both an inhaled corticosteriod and a long-acting beta 2 agonist.

The decision to prescribe fluticasone/formoterol fixed dose combination will precede and be independent of the decision to enroll the patient into the study

Exclusion Criteria:

* There are no specific exclusion criteria as this is an observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible to be prescribed fluticasone/formoterol fixed dose combination as follows:
  Patients not adequately controlled in inhaled corticosteriods and "as required" inhaled short acting beta 2 agonist or patients already adequately controlled on both an inhaled corticosteriod and a long-acting beta 2 agonist.
  The decision to prescribe fluticasone/formoterol fixed dose combination will precede and be independent of the decision to enroll the patient into the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Estimated); Primary Completion 2016-12-15 (Estimated); Study Completion 2016-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of frequency of spacer use on asthma control in patients in normal clinical practice | This measurement will be taken after 12 weeks of treatment
  the Asthma Control Questionnaire will be completed by subjects at study baseline and then after 12 weeks of treatment. Difference between the 2 will be the primary endpoint.

IPD SHARING:
Plan to Share IPD: Undecided